CLINICAL TRIAL: NCT02076685
Title: The Application of the N-acetyltransferase 2 (NAT2) Genotyping in Re-challenge Protocol of Isoniazid (INH) Titration in Patients With Anti-TB Medications-induced Hepatitis
Brief Title: NAT2 Genotyping in Re-challenge Protocol of INH Titration in Patients With Anti-TB Medications-induced Hepatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 200805015M
Record Dates: First submitted 2012-11-16; First posted 2014-03-03 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Hepatotoxicity
Keywords: pharmacogenetics; anti-tuberculosis drug; genetic polymorphism; isoniazid
MeSH Terms: interventions — Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- isoniazid rechalleng (Experimental): When patients encountered hepatotoxicity during the anti-TB treatment, genotyping and pk study of INH would be performed and dose adjustment accordingly.
  Interventions: Drug: isoniazid

INTERVENTIONS:
Drug: isoniazid — dose adjustment according to the pharmacogenomic results
  Other Names: Duracin, Rifina

SUMMARY:
To improve the treatment outcome in patients with tuberculosis and integrate the pharmacogenetics into clinical practice, the information of NAT2 genotyping was used in re-challenge protocol for isoniazid (INH) titration in patients with anti-tuberculosis medication-induced hepatitis.

ELIGIBILITY:
Inclusion Criteria:

1. >= 18 years.
2. Take INH for at least a week.
3. abnormal liver function (ALT (alanine, transaminase) increased by more than three times the upper limit of normal, or ALT higher than twice the upper limit of normal and total bilirubin higher than 2.0 mg / dL

Exclusion Criteria:

1.Taking INH before liver function abnormalities. 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-11; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
successful re-use of isoniazid for TB treatment | 6 months
  In this study, we would like to test the hypothesis of NAT2 genotyping helping in isoniazid rechallenge after patients experienced adverse effects of anti-TB treatment. Therefore, to observe the patients can re-use isoniazid successfully is an important outcome measure in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Shen Li Jiuan, Ph.D, Principal Investigator — Nationa Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan